CLINICAL TRIAL: NCT03395470
Title: A Double-blind, Randomised, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Doses of PXL770, Including an Open-label, One-sequence Part to Assess the Drug-drug Interaction With Rosuvastatin in Healthy Male Subjects
Brief Title: Safety, Tolerability and PK of PXL770 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poxel SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PXL770-002
Record Dates: First submitted 2017-11-06; First posted 2018-01-10 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases | interventions — 2-chloro-3-(1-hydroxy-5,6,7,8-tetrahydronaphthalen-2-yl)-6-oxo-5-phenyl-7H-thieno)(2,3-b)pyridin-4-olate potassium; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A1 (Experimental): Dose 1 or placebo
  Interventions: Drug: PXL770; Drug: Placebo
- Group A2 (Experimental): Dose 2 or placebo
  Interventions: Drug: PXL770; Drug: Placebo
- Group A3 (Experimental): Dose 3 or placebo
  Interventions: Drug: PXL770; Drug: Placebo
- Group A4 (Experimental): Dose 4 or placebo
  Interventions: Drug: PXL770; Drug: Placebo
- Group A5 (Experimental): Dose 5 or placebo
  Interventions: Drug: PXL770; Drug: Placebo
- Group B (Experimental): Dose + Rosuvastatin
  Interventions: Drug: PXL770; Drug: Rosuvastatin

INTERVENTIONS:
Drug: PXL770 — MAD
Drug: Placebo — MAD
  Arms: Group A1; Group A2; Group A3; Group A4; Group A5
Drug: Rosuvastatin — DDI
  Arms: Group B

SUMMARY:
PXL770 is a direct activator of 5' adenosine monophosphate-activated protein kinase (AMPK) being developed by Poxel S.A. for the treatment of type 2 diabetes mellitus (T2DM). In Part A of this study, we'll test the safety, tolerability and pharmacokinetics (PK) of repeated doses. In Part B, we'll co-administer PXL770 and rosuvastatin (a HMG-CoA reductase inhibitor) to assess any drug-drug interaction.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects deemed healthy on the basis of a clinical history, physical examination, ECG, vital signs, and laboratory tests of blood and urine
* body mass index in the range 18.5-29.9 kg/m²
* body weight at least 60 kg
* willing to use reliable contraception
* able to give fully informed written consent.

Exclusion Criteria:

* Pregnant or lactating woman, or sexually active woman of child-bearing potential not using reliable contraception
* Clinically relevant abnormal findings at the screening assessment
* Clinically significant vital signs outside the acceptable range at screening
* Clinically relevant abnormal medical history, surgery or concurrent medical condition
* Acute or chronic illness
* Estimated glomerular filtration rate less than 80 mL/min/1.73 m2
* Severe adverse reaction to any drug or sensitivity to the trial medication or its components
* Significant food allergy; vegetarian or vegan
* Participation in other clinical trials of unlicensed or prescription medicines, or loss of more than 400 mL blood, within the 3 months before first dose of trial medication
* Drug or alcohol abuse
* Smoking of more than 5 cigarettes daily
* Possibility that subject will not cooperate
* Positive test for hepatitis B & C, HIV
* Objection by a General Practitioner

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Part A: PK parameters of PXL770 after repeated doses Part B: PK parameters of rosuvastatin before and after repeated doses of PXl770 | From baseline to day 14
  - Cmax: peak plasma concentration after dosing
Part A: PK parameters of PXL770 after repeated doses | From baseline to day 14
  - AUC0-t: area under the concentration-time curve from 0 extrapolated to time t
Part A: PK parameters of PXL770 after repeated doses | From baseline to day 14
  - AUC0-∞: area under the concentration-time curve from 0 extrapolated to infinite

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From baseline to day 14
  Incidence of treatment emergent adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research (HMR), London, United Kingdom